CLINICAL TRIAL: NCT05129605
Title: Prostate Cancer Genetic Risk Evaluation and Screening Study (PROGRESS)
Brief Title: Prostate Cancer Genetic Risk Evaluation and Screening Study
Acronym: PROGRESS
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Keyan Salari, MD, PhD, Urologic Oncology, Massachusetts General Hospital
Other Study IDs: 2020P000081
Record Dates: First submitted 2021-11-02; First posted 2021-11-22 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Prostatic Neoplasm; Prostate Cancer; BRCA2 Mutation; BRCA1 Mutation; ATM Gene Mutation; MMR Mutation; Lynch Syndrome; Genetic Predisposition to Disease
Keywords: BRCA2; BRCA1; Mismatch Repair Deficiency; Lynch Syndrome; HOXB13; Family History of Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis; Genetic Predisposition to Disease; Turcot syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — * Blood and urine on all subjects
  * Tumor tissue on subjects who develop prostate cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort A: Documented germline known pathogenic or likely pathogenic mutation in a prostate cancer related risk gene
  Interventions: Diagnostic Test: Prostate cancer screening
- Cohort B: Family history suggestive of high genetic risk for prostate cancer with clinical genetic testing negative for known pathogenic or likely pathogenic mutations in prostate cancer-related risk genes
  Interventions: Diagnostic Test: Prostate cancer screening
- Cohort C: Individuals who self-identify as Black American or Black Caribbean with both parents and all four grandparents of Black/African ancestry
  Interventions: Diagnostic Test: Prostate cancer screening

INTERVENTIONS:
Diagnostic Test: Prostate cancer screening — Physical exam (digital rectal exam), prostate-specific antigen (PSA) and PSA derivatives, and multiparametric MRI of the prostate

SUMMARY:
This study aims to define the natural history of men at high genetic risk for prostate cancer on the basis of specific germline genetic mutations, family history, or Black/African ancestry and evaluate the utility of prostate MRI as a screening tool. The hypothesis is that this targeted population of men are at elevated risk of developing prostate cancer compared to the general population, and enhanced screening with MRI will enable early detection and diagnosis of potentially aggressive prostate cancer, characterization of the penetrance of specific mutations, and potentially identify new genetic risk mutations.

DETAILED DESCRIPTION:
Prostate cancer is the most common malignancy and the second leading cause of cancer-related deaths in American men. Prostate cancer has substantial inherited predisposition and men harboring specific genetic variants or a positive family history have been associated with an increased risk of developing prostate cancer. Men with specific genetic variants, such as pathogenic BRCA2 mutations, are at particularly greater risk of developing aggressive forms of prostate cancer and thus warrant undergoing careful screening for prostate cancer. However, the penetrance of many mutations in prostate cancer risk genes is unknown, and some men have no identifiable mutations in known risk genes despite a strong family history of prostate cancer. Prospectively collected clinical data along with biospecimens from unaffected individuals at high genetic risk for developing prostate cancer will advance the understanding of how specific mutations contribute to the development of prostate cancer and how these prostate cancers might be best detected. The purpose of this study is to prospectively screen men at high risk genetic risk for prostate cancer by prostate exam, PSA, and prostate MRI to characterize the penetrance and cancer-related outcomes of specific mutations, identify potentially novel genetic risk mutations and/or markers for early detection.

ELIGIBILITY:
Inclusion Criteria:

* Men 35-74 years old
* No known diagnosis of prostate cancer
* Life expectancy >10 years
* Meet cohort A, B, or C criteria
* Cohort A: Documented pathogenic or likely pathogenic germline genetic mutation in a prostate cancer risk gene from a CLIA-certified laboratory (ATM, ATR, BRCA1, BRCA2, BRIP1, CHEK2, EPCAM, FANCA, GEN1, HOXB13, MLH1, MSH2, MSH6, NBN, PALB2, PMS2, RAD51C, RAD51D, TP53)
* Cohort B: A strong family history suggestive of high genetic risk for prostate cancer with negative clinical genetic testing
* Cohort C: Individuals who self-identify as Black American or Black Caribbean with both parents and all four grandparents of Black/African ancestry

Exclusion Criteria:

* Prior diagnosis or treatment of prostate cancer
* Inability to undergo prostate MRI
* Inability to receive MRI contrast agent

Ages: 35 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men ages 35-74 years old at high genetic risk for prostate cancer on the basis of a specific germline genetic mutation or a strong family history.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of prostate cancer | From date of enrollment until date of diagnosis of prostate cancer or age of 75 reached, which ever came first
  Diagnosis of overall and clinically significant (grade group 2 or higher) prostate cancer

SECONDARY OUTCOMES:
Positive predictive value of multiparametric MRI for detection of prostate cancer | From date of enrollment until date of diagnosis of prostate cancer or age of 75 reached, which ever came first
  Positive predictive value of multiparametric prostate MRI for detecting clinically significant prostate cancer in men at high genetic risk for prostate cancer with a positive MRI (PI-RADS score of 3 or higher)

CONTACTS AND LOCATIONS:
Overall Officials: Keyan Salari, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amini AE, Salari K. Incorporating Genetic Risk Into Prostate Cancer Care: Implications for Early Detection and Precision Oncology. JCO Precis Oncol. 2024 Feb;8:e2300560. doi: 10.1200/PO.23.00560. PMID 38412389
- [Background] Amini AE, Hunter AE, Almashad A, Feng AJ, Patel ND, O'Dea MR, McCormick SR, Rodgers LH, Salari K. Magnetic Resonance Imaging-based Prostate Cancer Screening in Carriers of Pathogenic Germline Mutations: Interim Results from the Initial Screening Round of the Prostate Cancer Genetic Risk Evaluation and Screening Study. Eur Urol Oncol. 2024 Dec;7(6):1358-1366. doi: 10.1016/j.euo.2024.01.015. Epub 2024 Mar 6. PMID 38453598